CLINICAL TRIAL: NCT02953145
Title: The Use of Fibrin Sealant to Reduce Post Operative Pain in Cleft Palate Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of support
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45664
Record Dates: First submitted 2015-09-18; First posted 2016-11-02 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2021-09

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tisseel applied (Experimental): In this group, the fibrin sealant Tisseel will be applied as a hemostasis agent in patients undergoing primary palatoplasty
  Interventions: Drug: Tisseel
- No fibrin sealant (No Intervention): In this group, no fibrin sealant will be applied intra-operatively. Standard measures, such as electrocautery, will be used for hemostasis.

INTERVENTIONS:
Drug: Tisseel — Tisseel will be applied to open areas lateral to the cleft palate repair
  Other Names: fibrin sealant
  Arms: Tisseel applied

SUMMARY:
Cleft Palate is a condition which affects up to 1 in 500 live births. Current treatment is surgery to correct the underlying anomaly. Children born with cleft palate typically undergo surgery at age 12 months. Standard ways to stop surgical bleeding include direct pressure and the use of electrocautery (burning of the tissue). Other products are available to help lessen blood loss. One of these includes a fibrin sealant. Fibrin is the key component of a blood clot. When a fibrin sealant is applied there are a variety of potential benefits other than bleeding control. One of these is decreased pain post operatively It is the investigators belief that the use of a fibrin sealant, Tisseel, in cleft palate surgery will decrease pain and enhance the recovery of children who undergo cleft palate repair.

The proposed study will randomly select children undergoing cleft palate repair to have tisseel used on the incision. Through statistical tests 40 children will be recruited (20 to have tisseel used and 20 with no tisseel). The use of tisseel will be known to the surgeon but not to the recovery room or ward nursing staff. Post operatively, the FLACC pain scale will be used to score the pain of the children throughout their admission to the Stollery children's hospital. The amount of pain controlling medication required as well as time to discharge will also be recorded. Statistical analysis of the data will be performed using accepted methods. Overall, the investigators hope to show that fibrin sealant, tisseel, will less the amount of post operative pain experienced by children undergoing cleft palate repair.

DETAILED DESCRIPTION:
Cleft palate is a condition which affects up to 1:500 births. Current practice is that children are enrolled in a multidisciplinary care team and undergo primary cleft palate repair at 12 months of age. These children are admitted to hospital overnight for observation of airway compromise, bleeding and analgesics. The use of fibrin sealant is gaining popularity and its use in pediatric surgery is becoming more commonplace. It acts as both a hemostatic agent as well as an adhesive. A review of the current literature on fibrin sealant has shown that in adults and children it may decrease post operative inflammation and pain. In 1994 Moralee et al published that the use of fibrin sealant in tonsillectomy patients in lieu of diathermy resulted in decreased pain in the early post operative period and that it was equally effective as a hemostatic method. Another study published in 2005 by healy et al showed that when fibrin sealant was applied to the donor site from a thigh split thickness skin graft patients experienced significantly less pain over a 14 day study period. Tisseel is a safe product when used appropriately. It is contraindicated for injection intra-arterially and in those with allergy. It is derived from plasma however viral transmission has not been shown to occur in this product. A full product monograph is available. It is the investigators hypothesis that the use of tisseel in pediatric patients undergoing cleft palate repair will result in decreased post operative pain.

The proposed study is a prospective randomized control trial. The control group will have electrocautery as the primary method of hemostasis control and the treatment group will have tisseel applied to the incision. The primary outcome of the study is post operative pain. Secondary outcomes will be the amount of analgesics required during the hospital admission, time to discharge, time to first feeding, minor complication rates- infection, dehiscence, respiratory compromise, and long term sequelae- oronasal fistula formation, need for revision, velopharyngeal insufficiency. Statistical calculations for sample size have determined that 16 patients will be needed in each group. This was calculated based on an alpha of 0.05 and power(beta) of 0.8. Statistical significance will be set as p<0.05.

Recruitment will be directed at parents/guardians of patients to undergo cleft palate repair. Details of the study will be explained to parents pre-operatively. Currently the pediatric plastic surgeons at the Stollery Children's Hospital use tisseel in their repair techniques however the investigators do not have concrete data suggesting it has a clear benefit for this procedure. Two surgeons will be enrolling patients and performing surgeries independently with or without the assistance of residents and/or medical students. After informed consent by the primary decision maker, the patient will be randomized, via concealed envelop, to have Tisseel used or have electrocautery used as a hemostatic mechanism. The parents/guardians will be blinded to the randomization. The operating room staff will know the results of the randomization and will need to prepare the Tisseel product. All other health care providers caring for the patient in the recovery period will be blinded to the randomization. Post-operative pain scores will be determined using the FLACC (Face, Legs, Activity, Cry, Consolability) scoring system. This system is a validated objective pain scoring system used in young children post procedure. Patients will be assessed in the standard fashion. Pain scores and analgesic medications given will be recorded as per current nursing policy as well as on the study record which will be placed in the patient's chart. Parents will be shown how to assess FLACC scores and if patient is discharged prior to 72 hours, the parent or guardian will be asked to record the FLACC score at certain time points. The record of time to first feeding will be recorded on the study record form. Patients will be discharged from hospital when current criteria for safe discharge are met. Clinic follow up will be conducted in the current standard method at the surgeon's discretion. It will be noted on the patient's hospital chart that they were enrolled in this study in order to track long-term outcomes listed above.

Student t-test will be used to compare the outcome data. Demographic parameters will be collected to validate the randomization of the study groups. Age at time of surgery, associated congenital malformations including cleft lip and prior orthodontic surgery/interventions will be recorded and stored in a password protected data storage device. Results of the study will be made available to the parent/guardians of the study patients. It is estimated that the study will require one year of recruitment and data collection for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary cleft palate repair (palatoplasty)
* Informed consent from parent(s) or guardian(s)

Exclusion Criteria:

* Allergy to any component of Tisseel
* failure to obtain informed consent

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | time 1 hour post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 2 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 4 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 6 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 12 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 24 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 48 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.
Post operative pain | time 72 hours post operation
  FLACC scores will be determined by blinded ward nurses and/or caregiver of the patient.

SECONDARY OUTCOMES:
Requirement for analgesia | From immediate post operative period up to 5 days
  Any analgesic given to the patient will be recorded and compared for the two groups.
Time to discharge | From immediate post operative period up to 5 days
  Patients are discharged from hospital when they are feeding adequately, pain is controlled and there are no other complications. The time when the patient meets discharge criteria as well as the time they actually leave the ward will be recorded and assessed in this study.
Time to first feeding | From immediate post operative period up to 5 days
  The time to successful feeding can be used as a marker for tolerable pain post operatively. The time when the patient first feeds successfully will be recorded and compared for the two groups.
oronasal fistula | Immediately post operatively until 2 years post operatively.
  Patients will be followed in the cleft lip and palate clinic . For the two years post operatively, repaired cleft palates will be examined for the presence of oronasal fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Jaret L Olson, MD FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Stollery Alberta Children's hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis BR, Sandor GK. Use of fibrin glue in maxillofacial surgery. J Otolaryngol. 1998 Apr;27(2):107-12. PMID 9572465
- [Background] Healy C, Greig AVH, Murphy AD, Powell C, Pinder RJ, Saour S, Abela C, Knight W, Geh JLC. Prospective randomized controlled trial: fibrin sealant reduces split skin graft donor-site pain. Plast Reconstr Surg. 2013 Jul;132(1):139e-146e. doi: 10.1097/PRS.0b013e318299c6f4. PMID 23806933
- [Background] MacGillivray TE. Fibrin sealants and glues. J Card Surg. 2003 Nov-Dec;18(6):480-5. doi: 10.1046/j.0886-0440.2003.02073.x. PMID 14992096
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Moralee SJ, Carney AS, Cash MP, Murray JA. The effect of fibrin sealant haemostasis on post-operative pain in tonsillectomy. Clin Otolaryngol Allied Sci. 1994 Dec;19(6):526-8. doi: 10.1111/j.1365-2273.1994.tb01282.x. PMID 7895385